CLINICAL TRIAL: NCT06786572
Title: Interoceptive Training Enhanced Mindfulness (ITEM): Acceptability and Measurement
Brief Title: Interoceptive Training Enhanced Mindfulness
Acronym: ITEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H230149; 1R34AT012499-01A1 (NIH)
Record Dates: First submitted 2025-01-06; First posted 2025-01-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-11

CONDITIONS: Anxiety Sensitivity
Keywords: anxiety sensitivity; mindfulness; interoception

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interoceptive Training Enhanced Mindfulness (ITEM) (Experimental): Brief mindfulness training focused on management of unwanted internal sensations
  Interventions: Other: Mindfulness training
- Interoceptive Exposure (IE) (Active Comparator): Cognitive behavioral intervention featuring systematic exposure to unwanted internal sensations
  Interventions: Behavioral: Interoceptive exposure

INTERVENTIONS:
Other: Mindfulness training — Brief mindfulness training focused on management of unwanted internal sensations
  Arms: Interoceptive Training Enhanced Mindfulness (ITEM)
Behavioral: Interoceptive exposure — Cognitive behavioral therapy focused in interoceptive exposure to unwanted internal sensations
  Arms: Interoceptive Exposure (IE)

SUMMARY:
This pilot randomized controlled trial will compare a novel mindfulness training to interoceptive exposure to establish feasibility and acceptability as an intervention for anxiety sensitivity.

DETAILED DESCRIPTION:
Anxiety sensitivity (AS), which involves fear that arousal related symptoms will have negative physical, social or psychological ramifications, is an important driver of anxiety, trauma-related and somatic disorders. Cognitive behavioral therapy (CBT), particularly involving interoceptive exposure (IE; i.e., exposure to unwanted internal sensations), has the greatest demonstrated efficacy at reducing AS but can be hard to tolerate. Conversely, mindfulness is sought out for management of multiple mental health problems, but the observed clinical effects are often modest. A hybrid of these two approaches may capitalize on the strengths of each approach. Mindfulness training (MT) may increase the tolerability of exposure, enhance compliance and support extinction learning through increased engagement with the feared stimulus and heightened awareness of the nonoccurrence of feared outcomes. This project will evaluate the feasibility and acceptability of a novel hybrid intervention, Interoceptive Training Enhanced Mindfulness (ITEM), which combines IE with MT, evaluate its feasibility and acceptability. Forty-eight Veterans will be randomized to receive ITEM or IE in six one-on-one sessions delivered via telehealth. They will complete assessments before and after the 6-week intervention period. Outcomes related to engagement and compliance with ITEM and IE will be the primary focus. Because multiple mental health (e.g., anxiety, posttraumatic stress disorder, eating disorders and depression) and physical health (e.g., chronic pain, conditions related to toxic exposure) problems are driven by maladaptive reactions to interoceptive cues, this intervention has the potential to ultimately produce wide-spread mental and physical health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status
* able to read and speak English
* ASI-3 score of 23 or higher
* clinically meaningful distress/impairment related to an emotional or somatic complaint as determined by a Clinical Global Impression Scale (CGI) of 3 or greater
* Internet access via a device that can support remote study activities and ability to attend in person appointments

Exclusion Criteria:

* serious mental illness, including bipolar disorder or psychotic illness
* current, untreated alcohol or substance use disorder
* moderate-severe suicidality that would likely result in the need for urgent intervention in the next 2 months
* current regular meditation practice or treatment for AS-related condition
* cognitive dysfunction that interferes with the ability to engage in treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate | Typically up to 3 months, from initial referral to decision to enroll or not
  Number enrolled out of number approached
Attendance | During the six-week intervention period
  Average number of sessions attended
Clinician's judgment of proportion of completion of at home assignments | During the six-week intervention period
  Clinician's judgment of proportion of completion of at home assignments on a scale including none, partial and complete
Client Satisfaction Questionnaire-4 (CSQ-4) | Week 6, following the final treatment session
  The CSQ-4 is a validated measure of participant satisfaction with care delivered with higher scores (range 4-16) indicating greater satisfaction.
Reliable change | Over a 6-8 week period from baseline to post-treatment
  Proportion improved, unchanged and worsened based on the Reliable Change Index using the Overall Anxiety Symptoms and Impairment Scale (OASIS).

CONTACTS AND LOCATIONS:
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Final datasets in machine-readable format will be shared via PubMed Central
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available 3/31/28, indefinite
Access Criteria: Public access
URL: https://pmc.ncbi.nlm.nih.gov/